CLINICAL TRIAL: NCT06119048
Title: Phe for Me? A Precision Nutrition Clinical Trial of Metabolic, Cardiovascular, and Neurocognitive Responses to Phenylalanine Among Carriers and Non-carriers of PKU
Brief Title: Phe for Me? The Effects of L-Phe on PKU Carriers and Non-carriers
Acronym: Phe for Me
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: McMaster University (Other); Laval University (Other)
Responsible Party: Principal Investigator, Justine Keathley, Assistant Professor, University of Guelph
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-03-017
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Autosomal Recessive Disorder (Genetic Carriers of PKU)
MeSH Terms: interventions — Phenylalanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Genetic Carriers and Non-Carriers of PKU (Experimental)
  Interventions: Dietary Supplement: L-Phenylalanine

INTERVENTIONS:
Dietary Supplement: L-Phenylalanine — 100 mg/kg

SUMMARY:
This is a clinical intervention study of PKU carriers (cases) and non-carriers (controls). Upon completing the informed consent process, participants will complete baseline measures of chronic mental health prior to the intervention (PHQ-9, GAD-7, BIS-11). Participants will attend the Human Nutraceutical Research Unit (HNRU) at the University of Guelph, fasted, and first undergo baseline measures of cognition and acute mental health (mood) and provide samples or saliva, urine and dried blood spots to evaluate phenylalanine (Phe), tyrosine (Tyr) and their metabolites (PAH pathway functioning) as well as for genetic testing of the PAH gene. Participants will also complete a brief questionnaire which will include age, sex, ethnicity, income, weight and height (measured using a stadiometer and calibrated weigh scale), and confirmation that participants arrived to the lab fasted (i.e. have only had water to drink and no other foods/ beverages prior to analyses). Blood pressure and heart rate will also be measured at baseline.

Following baseline tests, participants will consume a pure L-Phe supplement dosed at 100 mg/kg mixed with 125 mL of water and 125mL of orange juice. Blood pressure and heart rate will be repeated at 1-hour post-L-Phe consumption. Two-hours postprandial, participants will repeat the cognitive tests and acute mental health (mood) assessment, blood pressure and heart rate measurement and provide follow-up saliva, urine and dried blood spot samples. Participants will also be asked to report any side effects they experienced with the L-Phe consumption.

ELIGIBILITY:
Inclusion Criteria:

* Carrier or non-carrier of PKU
* At least 18 Years of age
* Comfortable fasting the morning of the study (no food or drink other than water)

Exclusion Criteria:

* Diagnosed with: PKU, severe neurodegenerative conditions affecting cognition (e.g. Alzheimer's, Parkinson's, dementia), melanoma, hypertension, liver disease and/or kidney disease
* Diagnosed with hypertension or hypotension
* Taking a monoamine oxidase inhibitor anti-depressant
* Pregnant or breastfeeding
* Orange/citrus allergy or intolerance
* Body weight 150 kg or greater
* History of fainting during blood sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Stop Signal Reaction Time | Change from baseline to 2-hours post L-Phe supplementation
  Response Inhibition

SECONDARY OUTCOMES:
Working Memory | Change from baseline to 2-hours post L-Phe supplementation
  N-Back Test Outcome
Individual Coefficient of Variance (Variability in Reaction Time) | Change from baseline to 2-hours post L-Phe supplementation
  Stop Signal Task Outcome
Phenylalanine Levels | Change from baseline to 2-hours post L-Phe supplementation
  Blood, saliva and urine sample analyses
Tyrosine Levels | Change from baseline to 2-hours post L-Phe supplementation
  Blood, saliva and urine sample analyses
Phenylalanine Metabolites | Change from baseline to 2-hours post L-Phe supplementation
  e.g. phenylethylamine, tyramine, phenylpyruvate, others
Tyrosine Metabolites | Change from baseline to 2-hours post L-Phe supplementation
  e.g. L-DOPA, dopamine, norepinephrine, epinephrine, p-hydroxyphenylpyruvate, homogentisic acid, fumarate, others
Mood | Change from baseline to 2-hours post L-Phe supplementation
  Profile of Mood State (POMS) Outcome
Blood Pressure | Change from baseline to 1-hour and 2-hours post L-Phe supplementation
  Systolic and Diastolic
Heart rate | Change from baseline to 1-hour and 2-hours post L-Phe supplementation
  BPM
Side Effects Following L-Phe Consumption | 0-3 hours post L-Phe consumption
  To be monitored throughout the visit to the research unit

OTHER OUTCOMES:
Chronic Anxiety | Baseline
  GAD-7 Outcome (higher scores indicate worse anxiety: range of 0 to >15)
Chronic Depression | Baseline
  PHQ-9 Outcome (higher scores indicate worse depression: range of 0 to 27)
Impulsivity | Baseline
  BIS-11 Outcome (higher scores indicate more impulsivity: range 30 to 120)
Trial-by-Trial Analysis | Change from baseline to 2-hours post L-Phe supplementation
  to be conducted if there are significant findings from the four main stop signal task outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No